CLINICAL TRIAL: NCT01385839
Title: Efficacy of Hair Transplantation Compared With Hypodermic Needle Irritation in Alopecia Areata
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-0533
Record Dates: First submitted 2011-06-28; First posted 2011-06-30 (Estimated); Last update posted 2016-12-22 (Estimated); Status verified 2016-12

CONDITIONS: Alopecia Areata; Alopecia; Balding
Keywords: Alopecia; Hair transplantation; Needle irritation; Medical needling
MeSH Terms: conditions — Alopecia Areata; Alopecia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- alopecia areata (Experimental): pts will have one area (or ½ of a large area) treated by hair transplant and another (or the other ½) treated by simple irritation with a large gauge sterile hypodermic needle
  Interventions: Procedure: Hair transplantation; Procedure: Hypodermic needle irritation

INTERVENTIONS:
Procedure: Hair transplantation — Hair transplantation is a procedure in which donor hair follicles are harvested from a section of a patient's scalp, and transplanted in another bald recipient area, at which time it will take root and continue to grow. Hairs generally continue to grow indefinitely.Hair transplant involves mild sedation with Valium, followed by local anesthesia of the donor and recipient areas. Donor hair is harvested using a scalpel to cut narrow strips of hair bearing areas. Follicular units are obtained by slicing the donor tissue into naturally occurring groupings. The follicular units are placed into holes made by a hypodermic needle in the alopecia areata affected areas of the subject. Grafts are held in place by coagulated blood. A bandage is applied after the procedure and left in place over night. The following day, the patient returns for follow up, bandage removal, cleansing, hair washing, and a check up.
Procedure: Hypodermic needle irritation — In the areas which are simply treated with irritation with the hypodermic needle, the procedure is the same, except no follicular units are placed into the holes.

SUMMARY:
The purpose of this study is to look at the safety, as well as the efficacy of hair transplantation compared with irritation with hypodermic needles in the treatment of subjects with refractory alopecia areata.

With this study, the investigators hope to demonstrate that trauma is just as effective as hair transplant in the treatment of recalcitrant alopecia areata of the scalp.

DETAILED DESCRIPTION:
Alopecia areata is a recurrent, non-scarring type of hair loss that can affect any hair-bearing area. This disorder can present in many different manners. Though medically benign, alopecia areata can result in severe emotional and psychosocial stress in affected individuals. This disease can be treated by hair transplantation.

Hair transplantation is a procedure in which donor hair follicles are harvested from a section of a patient's scalp, and transplanted in another bald recipient area, at which time it will take root and continue to grow. Hairs generally continue to grow indefinitely

During this study, subjects with alopecia areata will have one area (or ½ of a large area) treated by hair transplant and another (or the other ½) treated by simple irritation with a large gauge sterile hypodermic needle.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must have recalcitrant, quiescent, alopecia areata, non-responsive to treatment, for at least 6 months.
2. Subject must have one patch of alopecia areata greater than 5 cm diameter, of two patches of alopecia areata, each greater than 2.5 cm diameter.

Exclusion Criteria:

1. Subjects with active, progressive, alopecia areata.
2. Subjects who are actively experiencing significant spontaneous regrowth of terminal hair.
3. Subjects with autoimmune deficiency.
4. Subjects with a medical condition contraindicating use of anesthesia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2009-10; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Change in follicular growth | day 0
  The study will require 5 study visits: Day 0, Day 1, Week 2, Week 24, and Week 36.
Change in follicular growth | day 1
  The study will require 5 study visits: Day 0, Day 1, Week 2, Week 24, and Week 36.
Change in follicular growth | 2 weeks
  The study will require 5 study visits: Day 0, Day 1, Week 2, Week 24, and Week 36.
Change in follicular growth | 24 weeks
  The study will require 5 study visits: Day 0, Day 1, Week 2, Week 24, and Week 36.
Change in follicular growth | 36 weeks
  The study will require 5 study visits: Day 0, Day 1, Week 2, Week 24, and Week 36.

CONTACTS AND LOCATIONS:
Overall Officials: Robin Unger, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, Department of Dermatology Clinical Trials Center, New York, New York, United States

REFERENCES:
- [Background] Civas E, Aksoy B, Aksoy HM, Eski M, Yucel K. Hair transplantation for therapy-resistant alopecia areata of the eyebrows: is it the right choice? J Dermatol. 2010 Sep;37(9):823-6. doi: 10.1111/j.1346-8138.2010.00872.x. PMID 20883369
- [Background] Barankin B, Taher M, Wasel N. Successful hair transplant of eyebrow alopecia areata. J Cutan Med Surg. 2005 Aug;9(4):162-4. doi: 10.1007/s10227-005-0136-x. PMID 16502201
- [Background] Delamere FM, Sladden MM, Dobbins HM, Leonardi-Bee J. Interventions for alopecia areata. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD004413. doi: 10.1002/14651858.CD004413.pub2. PMID 18425901
- [Background] Garg S, Messenger AG. Alopecia areata: evidence-based treatments. Semin Cutan Med Surg. 2009 Mar;28(1):15-8. doi: 10.1016/j.sder.2008.12.002. PMID 19341938
- [Background] Lee JW, Yoo KH, Kim BJ, Kim MN. Photodynamic therapy with methyl 5-aminolevulinate acid combined with microneedle treatment in patients with extensive alopecia areata. Clin Exp Dermatol. 2010 Jul;35(5):548-9. doi: 10.1111/j.1365-2230.2009.03695.x. Epub 2009 Nov 3. No abstract available. PMID 19886963